CLINICAL TRIAL: NCT02116257
Title: The Opioid-sparing Effect and Reduced PONV Using Propacetamol in PCA Among Patients With High Risk of PONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2013-0702
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: PONV; Propacetamol
Keywords: Nausea; Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — propacetamol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propacetamol (Experimental)
  Interventions: Drug: Propacetamol
- PCA regimen (Placebo Comparator): routine PCA drug
  Interventions: Drug: PCA regimen

INTERVENTIONS:
Drug: Propacetamol — total 4g of Propacetamol added to patient's PCA regimen
  Arms: Propacetamol
Drug: PCA regimen
  Arms: PCA regimen

SUMMARY:
While Patient-controlled analgesia (PCA) has the advantage of effectively reducing the degree of postoperative pain, it can also affect the patient's outcome by several adverse effects such as postoperative nausea and vomiting (PONV). Especially for high risk group of patients for PONV, the ideal regimen for sufficient analgesia with minimal adverse effect needs to be sought. Propacetamol is known for its effective, rapid analgesia, opioid-sparing effect, and is used widely for post operative pain management. This study aims to see the opioid-sparing effect and the degree of PONV when propacetamol is added to PCA for high risk PONV patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for either 1-2 level spine fusion or laminectomy
2. ASA (American Society of Anesthesiology) physical status 1 or 2
3. Non-smoking female patients, between the age 20 and 65

Exclusion Criteria:

1. Administration of any anti-emetic agents within 24 hours prior to surgery
2. Administration of any opioid agents within 7 days prior to surgery
3. Regular administration of any steroid agents
4. Drug or alcohol-abuser
5. Patients with bowel movement disorder, liver or renal impairment, insulin-dependent diabetes. Patients who are pregnant, illiterate, or foreign.
6. Patients administered to Intensive Care Unit after surgery

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence of PONV | from immediate postop to 24 hours after the surgery
  Incidence of postoperative nausea, vomiting - Number of events

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea